CLINICAL TRIAL: NCT04979442
Title: A Randomized Multicenter Phase 3 Study of Milademetan Versus Trabectedin in Patients With Dedifferentiated Liposarcoma
Brief Title: Treatment of Milademetan Versus Trabectedin in Patient With Dedifferentiated Liposarcoma
Acronym: MANTRA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAIN-3201
Record Dates: First submitted 2021-07-06; First posted 2021-07-28 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Dedifferentiated Liposarcoma
Keywords: sarcoma; MDM2; pleomorphic liposarcoma
MeSH Terms: conditions — Liposarcoma; Sarcoma | interventions — milademetan; Trabectedin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RAIN-32 (Milademetan) (Experimental): 260 mg once daily orally on Days 1 to 3 and Days 15 to 17 of each 28-day cycle.
  Interventions: Drug: RAIN-32
- Trabectedin (Active Comparator): 1.5 mg/m2 body surface area as a 24-hour IV infusion, every 3 weeks.
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: RAIN-32 — 260 mg once daily orally on Days 1 to 3 and Days 15 to 17 of each 28-day cycle
  Other Names: Milademetan
  Arms: RAIN-32 (Milademetan)
Drug: Trabectedin — 1.5 mg/m2 body surface area as a 24-hour IV infusion, every 3 weeks
  Other Names: Yondelis
  Arms: Trabectedin

SUMMARY:
Randomized, multicenter, open-label, Phase 3 registration study designed to evaluate the safety and efficacy of milademetan compared to trabectedin in patients with unresectable (i.e., where resection is deemed to cause unacceptable morbidity or mortality) or metastatic DD liposarcoma that progressed on 1 or more prior systemic therapies, including at least 1 anthracycline-based therapy.

DETAILED DESCRIPTION:
Approximately 160 patients will be randomly assigned in a 1:1 ratio to receive milademetan or trabectedin. Randomization will be stratified by the ECOG performance status (0 or 1) and number of prior treatments (≤ 2 or > 2) for the patient's liposarcoma.

Patients will receive study drug (i.e., milademetan or trabectedin) until reaching unequivocal disease progression (RECIST v.1.1) as determined by the Investigator, experiencing unmanageable toxicity, or until other treatment discontinuation criteria are met. Patients may be treated beyond tumor progression if they are experiencing clinical benefit based on the assessment of the Investigator in discussion with the Medical Monitor. All patients will be followed for documentation of disease progression and survival information (i.e., date and cause of death) and subsequent treatment information (i.e., date/duration of treatment, response, and subsequent disease progression). Long-term follow-up will continue every 12 weeks (± 7 days) until the endpoint of death, the patient is lost to follow-up, or for 24 months following the final dose of study drug, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DD liposarcoma, with or without a WD component (WD/DD liposarcoma). Note: Patient must be willing to provide an archival tumor tissue sample that is ≤ 3 years old and of adequate quality or willing to provide a fresh pretreatment biopsy sample
* Advanced unresectable (i.e., where resection is deemed to cause unacceptable morbidity or mortality) and/or metastatic WD/DD liposarcoma
* Measurable tumor lesion(s) in accordance with RECIST version 1.1
* Received 1 or more systemic cancer therapy regimens, including at least 1 anthracycline-based regimen, and had radiographic progressive disease (per RECIST version 1.1) within 6 months before the Screening Visit
* Resolution of any clinically relevant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy
* ECOG performance status of 0 or 1
* Adequate bone marrow function:

  * Platelet count ≥ 100 × 10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1.5 × 10^9/L
* Adequate hepatic function:

  * Alanine aminotransferase and aspartate aminotransferase ≤ 3 × upper limit of normal (ULN) if no liver metastases are present; ≤ 5 × ULN if liver metastases are present
  * Total bilirubin ≤ 1.5 × ULN, or ≤ 3 x ULN in the setting of Gilbert's disease

Exclusion Criteria:

* Prior treatment with any mouse double minute 2 (MDM2) inhibitor or trabectedin
* Other primary malignancies that have required systemic antineoplastic treatment within the previous 2 years, except for localized cancers that have apparently been cured
* Gastrointestinal conditions that could affect the absorption of milademetan, in the opinion of the Investigator
* Uncontrolled infection within the last 7 days requiring IV antibiotics, antivirals, or antifungals
* Known HIV infection or active Hepatitis B or C
* Untreated brain metastases. Note: Patients who require steroids for brain metastases must be on a stable or tapering dose of corticosteroids for at least 2 weeks before randomization. If applicable, patients must complete stereotactic radiosurgery 7 days before and whole brain radiotherapy 21 days before their first dose of study drug.
* Investigational therapy administered within the 28 days or 5 half lives:

  1. Cytochrome P450 3A4 isozyme strong inhibitor: 5 elimination half-lives
  2. CYP3A strong or moderate inducers: 4 weeks
  3. Systemic anticancer therapy or investigational therapy 3 weeks or 5 half-lives,
  4. Immunotherapy with checkpoint inhibitor: 4 weeks
* Curative-intent radiation therapy ≤ 4 weeks or palliative radiation therapy,
* Uncontrolled or significant cardiovascular disease:

  1. QTcF at rest, where the mean QTcF interval is > 480 milliseconds
  2. Myocardial infarction within 6 months
  3. Uncontrolled angina pectoris within 6 months
  4. New York Heart Association Class 3 or 4 congestive heart failure
  5. Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (22):
  - Stanford Cancer Center, Palo Alto, California
  - Sarcoma Oncology Research Center, LLC, Santa Monica, California
  - UCLA Department of Medicine - Hematology/ Oncology, Santa Monica, California
  - CU Anschutz Medical Campus, Anschutz Cancer Pavilion, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami Hospital & Clinics - Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago Heights, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University School of Medicine, Duke Cancer Institute, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Austria (3):
  - Order Hospital Linz - Sisters of Mercy, Linz
  - University Hospital Salzburg, Salzburg
  - Medical University Vienna, Department of Internal Medicine I, Vienna
- Belgium (2):
  - Ghent University, Oncology Center, Ghent
  - University Hospitals Leuven Campus Gasthuisberg, Leuven
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (9):
  - Georges-Francois Leclerc Cancer Research Center, Dijon, Bourgogne-Franche-Comté
  - ICANS, Strasbourg, Grand Est
  - Institut Bergonie, Bordeaux, Nouvelle-Aquitaine
  - Centre Hospitalier de Poitiers, Poitiers, Nouvelle-Aquitaine
  - Institute Claudius Regaud, Toulouse, Occitanie
  - Centre Antoine Lacassagne, Nice, Provence-Alpes-Côte d'Azur Region
  - CHU La Timone - Oncologie medicale, Marseille, Prvence-Alpes-Cote d'Azu
  - Leon Berard Center, Lyon
  - Gustave Roussy, Villejuif
- Georgia (5):
  - LTD High -Tech Hospital MedCenter, Batumi
  - LLC Todua Clinica, Tbilisi
  - LTD Health House, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicin Center LLC, Tbilisi
  - LTD Caucasus Medical Centre, Tbilisi
- Germany (6):
  - Helios Hospital Bad Saarow, Clinic for Hematology, Oncology and Palliative Medicine, Bad Saarow, Bradenburg
  - HELIOS Hospital Berlin-Buch, Berlin
  - University Medical Center-Mainz, Mainz
  - University Hospital Mannheim, Mannheim Cancer Center, Mannheim
  - Münster University Hospital, Münster
  - University Hospital Ulm, Ulm
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong
- St Vincent's University Hospital, Dublin, Ireland
- Italy (8):
  - National Cancer Institute, IRCCS, Milan
  - National Cancer Institute-IRCCS "Fondazione G. Pascale", Naples
  - Veneto Oncology Institute (IOV), IRCCS, Padua
  - University Polyclinic Hospital "Paolo Giaccone" Palermo, Palermo
  - Santo Stefano Hospital of Prato - USL Company Toscana Center, Prato
  - Santo Stefano Hospital - ASL 4 Toscana, Prato
  - University Hospital Campus Bio-Medico, Rome
  - Institute of Cancer Research and Treatment of Candiolo - IRCCS, Turin
- M. Curie National Research Institute of Oncology, Department of Soft Tissue/Bone Sarcoma and Melanoma, Warsaw, Poland
- South Korea (3):
  - Severance Hospital, Yonsei University Health System Seoul, Seoul
  - Asan Medical Center, Department of Oncology, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Passeig de la Vall d'Hebron 119-129, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - University General Hospital Gregorio Marañon, Madrid
  - University Hospital Foundation Jimenez Diaz, Madrid
  - University Hospital Miguel Servet, Zaragoza
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - The Royal Marsden Hospital NHS Foundation Trust, London, Chelsea
  - The Christie NHS Foundation Trust, Department of Medical Oncology, Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 86 subjects were enrolled to the Milademetan arm and a total of 89 subjects were enrolled to the Trabectedin arm. Of the 89 subjects in the trabectedin arm, 79 subjects were treated.
Groups:
- Milademetan: Milademetan was supplied as 30- and 100-mg strength capsules. The starting dose of milademetan 260 mg administered once daily (QD) orally on Days 1 to 3 and Days 15 to 17 of each 28-day cycle.
- Trabectedin: Trabectedin was provided as a sterilized lyophilized powder in single, 1-mg dose vials. Trabectedin was administered per the manufacturer's instructions at 1.5 mg/m2 body surface area (BSA) as a 24-hour IV infusion, every 3 weeks (ie, 21-day cycles) through a central venous line.
Period: Overall Study
Arm/Group | Milademetan | Trabectedin
Started | 86 | 89
Received Treatment | 86 | 79
Completed | 34 | 42
Not Completed | 52 | 47
Not completed — Death | 43 | 30
Not completed — Withdrawal by Subject | 8 | 13
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — do not want to continue | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Milademetan: milademetan 260 mg once daily orally on Days 1 to 3 and Days 15 to 17 of each 28-day cycle
- Trabectedin: trabectedin 1.5 mg/m2 body surface area as a 24-hour IV infusion, every 3 weeks
- Total: Total of all reporting groups
Arm/Group | Milademetan | Trabectedin | Total
Number analyzed (Participants) | 86 | 89 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.08) | 61.8 (11.92) | 60.6 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 76
  Male | 46 | 53 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 71 | 72 | 143
  Unknown or Not Reported | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 15 | 12 | 27
  Race: Black or African American | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: White | 59 | 63 | 122
  Race: Unknown | 11 | 12 | 23
  Race: Other | 0 | 0 | 0
Region [Count of Participants; unit: Participants]
  North America | 27 | 37 | 64
  Europe | 47 | 42 | 89
  Rest of World | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Compare Progression-free Survival (PFS) as Determined by Blinded Independent Central Review (BICR) Between the Milademetan Treatment Arm and Trabectedin Control Arm
Description: PFS is defined as the time from randomization to the earliest date of the first objective documentation of radiographic disease progression, or death due to any cause. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: from the randomization date to date of documented progression or death, up to 13 months
Population: Analysis population included all the randomized participants up to up to final analysis cut-off date (01 March 2023).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Milademetan | Trabectedin
Number analyzed (Participants) | 86 | 89
months | 3.6 [2.1 to 4.1] | 2.2 [1.9 to 4.2]

2. Secondary Outcome: Overall Survival (OS)
Description: OS as measured from the date of randomization to date of death by any cause
Time Frame: From randomization date to death. The result is based on primary analysis data cut.
Population: Analysis population included all the randomized participants up to up to final analysis cut-off date (01 March 2023).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Milademetan | Trabectedin
Number analyzed (Participants) | 86 | 89
months | 9.5 [6.5 to 12.8] | 10.2 [8.6 to NA] — Upper limit of the 95% confidence interval not estimable due to insufficient number of participants with events.

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR defined as the percentage of patients who have achieved CR, PR, or SD for >= 16 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From the randomization date to first CR, PR or SD >= 16 weeks or the primary study completion date; up to 26.6 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Milademetan | Trabectedin
Number analyzed (Participants) | 86 | 89
percentage of participants | 33.7 [23.9 to 44.7] | 27.0 [18.1 to 37.4]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR defined as the percentage of patients who have achieved a confirmed CR, PR. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From randomization date to the first confirmed complete or partial response, or study completion date; up to 26.6 months.
Population: This analysis is conducted in all participants within the Intent to treat (IIT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Milademetan | Trabectedin
Number analyzed (Participants) | 86 | 89
percentage of participants | 4.7 [1.3 to 11.5] | 3.4 [0.7 to 9.5]

5. Secondary Outcome: PFS by Investigator Assessments
Description: PFS defined as the time from randomization to the earliest date of the first objective documentation of radiographic disease progression or death due to any cause, based on Investigator assessments
Time Frame: disease progression or death
Population: PFS defined as the time from randomization to the earliest date of the first objective documentation of radiographic disease progression or death due to any cause, based on Investigator assessments
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Milademetan | Trabectedin
Number analyzed (Participants) | 86 | 89
months | 3.7 [2.1 to 5.4] | 2.1 [1.9 to 3.9]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Until Approximately 30 Days After the Last Study Drug
Description: All AEs were collected from the initiation of study treatment until 30 days after the last administration study drug or until initiation of another anticancer therapy, whichever came first; up to 26.6 months.
Time Frame: From first dose date to 30 days after the last dose date or the primary study completion date whichever came first; up to 26.6 months.
Population: All AEs were collected from the initiation of study treatment until 30 days after the last administration study drug or until initiation of another anticancer therapy, whichever came first.
Measure: Count of Participants; unit: Participants
Arm/Group | Milademetan | Trabectedin
Number analyzed (Participants) | 86 | 79
Participants | 86 | 78

ADVERSE EVENTS:
Time Frame: From the first dose date to 30 days after the last dose date or the primary study completion date whichever came first; up to 26.6 months.
Description: All-cause mortality assessed for all enrolled participants, serious and other adverse events assessed for safety population
Arm/Group | Milademetan | Trabectedin
All-Cause Mortality (participants affected / at risk) | 43/86 | 30/89
Serious Adverse Events (participants affected / at risk) | 31/86 | 38/79
Other Adverse Events (participants affected / at risk) | 86/86 | 78/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milademetan (N=86) | Trabectedin (N=79)
Anaemia (Blood and lymphatic system disorders) | 14 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 5
Sepsis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2
platelet count decreased (Investigations) | 3 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milademetan (N=86) | Trabectedin (N=79)
Nausea (Gastrointestinal disorders) | 61 | 46
Anemia (Blood and lymphatic system disorders) | 38 | 29
Vomiting (Gastrointestinal disorders) | 38 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 31 | 11
Fatigue (General disorders) | 30 | 26
Asthenia (General disorders) | 28 | 19
Decreased appetite (Metabolism and nutrition disorders) | 25 | 17
Diarrhea (Gastrointestinal disorders) | 24 | 21
platelet count decreased (Investigations) | 22 | 9
Neutrophil count decreased (Investigations) | 21 | 15
Abdominal pain (Gastrointestinal disorders) | 16 | 10
Neutropenia (Blood and lymphatic system disorders) | 15 | 14
Constipation (Gastrointestinal disorders) | 10 | 20
White blood cell count decreased (Investigations) | 12 | 8
Alanine aminotransferase increased (Investigations) | 4 | 20
Blood alkaline phosphatase increased (Investigations) | 4 | 12
Aspartate aminotransferase increased (Investigations) | 2 | 13
Acute kidney injury (Renal and urinary disorders) | 1 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Edema peripheral (General disorders) | 4 | 9
Blood creatinine increased (Investigations) | 8 | 7
Headache (Nervous system disorders) | 7 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 5
COVID-19 (Infections and infestations) | 7 | 6
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pyrexia (General disorders) | 3 | 6
Weight decreased (Investigations) | 3 | 4
Chills (General disorders) | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5
Mucosal inflammation (General disorders) | 2 | 4
Myalgia (General disorders) | 2 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 4
Gamma-glutamyl transferase increased (Investigations) | 0 | 7
Pain (General disorders) | 0 | 4
Lymphocyte count decreased (Investigations) | 3 | 5
Dysgeusia (Gastrointestinal disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT04979442/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT04979442/SAP_001.pdf